CLINICAL TRIAL: NCT04638153
Title: A PHASE 2 MULTIPLE DOSE, RANDOMIZED STUDY TO ASSESS THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND EFFICACY OF RECIFERCEPT IN CHILDREN WITH ACHONDROPLASIA
Brief Title: A Study Of Safety, Tolerability And Effectiveness Of Recifercept In Children With Achondroplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy at any of the tested doses on 18th November 2022. The decision to terminate the study is not related to a safety concern.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C4181005; 2020-001189-13 (EudraCT Number)
Record Dates: First submitted 2020-09-15; First posted 2020-11-20 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Achondroplasia
Keywords: Skeletal Dysplasia
MeSH Terms: conditions — Achondroplasia; Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Anthropometric Measurements Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Low Dose (Experimental): Low Dose
  Interventions: Biological: Recifercept
- Medium Dose (Experimental): Medium Dose
  Interventions: Biological: Recifercept
- High Dose (Experimental): High Dose
  Interventions: Biological: Recifercept
- PK Phase 2 Formulation (Experimental): Phase 2 formulation [process 1c] 3mg/kg
  Interventions: Biological: Recifercept
- PK Phase 3 Formulation (Experimental): Phase 3 formulation [process 2] 3mg/kg
  Interventions: Biological: Recifercept

INTERVENTIONS:
Biological: Recifercept — Recifercept

SUMMARY:
Approximately 63 participants will be randomized to one of three doses to receive Recifercept either

* Low Dose
* Medium Dose
* High Dose

Participants will will attend the clinic at baseline and at Day 1, 4, 8, 15, 29 & then Month 2, 3 6, 9 & 12. Assessments include safety, blood sampling, physical examination, vital signs, anthropometric body measurements & patient/caregiver quality of life questionnaires

Participants will received treatment with Recifercept for 12 months. All participants who complete the study and in the opinion of the investigator, continue to have a positive risk:benefit profile, will be offered to enroll into an open-label extension (OLE) study.

A PK cohort will include 12 participants who will randomly receive a single dose of 3 mg/kg of Phase 2 study (process 1c) formulation and a single dose of 3 mg/kg of the proposed Phase 3 (process 2) study formulation in a cross over study. Dose of the cohort could be changed due to emerging safety and efficacy data in the study.

DETAILED DESCRIPTION:
This is a phase 2 randomized, 3 arm (3 active doses of Recifercept), parallel group dose finding study of safety, tolerability, PK and efficacy

The total number of participants is 63 in 2 age straified cohorts of 0-2 years and 6-10 years old.

The study will enroll approximately 54 children with achondroplasia aged 2-10 years (inclusive) who will be enrolled and randomized to receive one of three doses of recifercept

* Low Dose
* Medium Dose
* High Dose

A total of 18 participants will be enrolled per dose 18 per dosesuch that at least 15 participants per dose are evaluable. An interim analysis is planned when at least 15 participants per dose aged ≥2 to <11 years have received 6 months of treatment with recifercept. eDMC will review safety, PK and efficacy data to confirm ongoing positive benefit:risk in participants.

Additionally, an exploratory cohort of approximately 9 children with achondroplasia, ages 0-2 years, will be enrolled later in the study (n=3 per dose).

Enrollment will follow an age and dose-staggered approach (descending age and ascending dose) with review of safety and PK data by the study team before progression to the next enrollment block If certain pre-defined safety signals occur then a meeting of the eDMC will be convened to make a decision on progression of enrollment. The PK data collected in block A will be used in the PopPK model (developed using healthy adult data) to confirm the dosing for younger children (ie, ≥2 to <6 years and 0-<2 years).

Participants will will attend the clinic at baseline and at Day 1, 4, 8, 15, 29 & then Month 2, 3 6, 9 & 12. Assessments include safety, blood sampling, physical examination, vital signs, anthropometric body measurements & patient/caregiver quality of life questionnaires

All participants will receive recifercept for 12 months. All participants who complete the study and in the opinion of the investigator, continue to have a positive risk:benefit profile, will be offered to enroll into an open-label extension (OLE) study.

PK Cohort:

Multiple changes have been made in the manufacturing process of the drug product (process 2) which will be used in Phase 3. Therefore, an additional PK cohort (at selected sites only) has been added, to evaluate the PK of Phase 2 formulation (process 1c) and Phase 3 formulation (process 2).

PK Cohort:

At selected sites only, an additional PK cohort has been added to evaluate the PK of two recifercept formulations. A total of 12 children with achondroplasia aged 2- <11 years will be enrolled in the PK cohort (6 in each treatment sequence). Each participant will receive 2 treatments (3 mg/kg Phase 2 formulation [process 1c] and 3 mg/kg Phase 3 formulation [process 2]) in a randomized manner. Dose of the cohort could be changed due to emerging safety and efficacy data in the study.

PK samples collected following each dose will be analyzed to evaluate the exposures of two formulations.

ELIGIBILITY:
Inclusion Criteria:

* Main cohort: Aged ≥2 years to <11 years (up to the day before 11th birthday inclusive) at time of enrollment; or exploratory cohort: aged ≥3 months to <2 years (up to the day before 2nd birthday inclusive) at time of enrollment
* Documented, confirmed genetic diagnosis of achondroplasia from historical medical records prior to entry into this trial (test must have been performed at a laboratory fully accredited for genetic testing under local regulations).
* Completed the C4181001 natural history study with at least 2 valid height/length measurements (at least 3 months apart) prior to enrollment in this study. One of these measurement timepoints must be within the 3 months prior to enrollment in C4181005.
* Tanner stage 1 based on investigator assessment during physical examination (must include assessment of breast development for females, testicular stage for males).
* Able to stand independently for height measurements (if ≥2 years of age at enrollment).
* If aged <2 years at enrollment, has a documented historical MRI brain/cervical spine performed in the previous 12 months.

Exclusion Criteria:

* Presence of co-morbid conditions or circumstances that, in the opinion of the investigator, would affect interpretation of growth data or ability to complete the trial procedures.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Presence of severe obesity (BMI >95th percentile on Hoover-Fong BMI charts) [Hoover-Fong et al, 2008].14
* Known closure of long bone growth plates (cessation of height growth).
* Body weight <7 kg or >30 kg.
* Moderate or severe renal impairment CrCL GFR <60 mL/min/1.73m2 (Calculated GFR based on updated "bedside" Schwartz formula for pediatric patients (CrCL (mL/min/1.73 m2) = 0.413 * Height (cms)/ Serum cr (mg/dL) or hepatic impairment (AST/ALT >1.5 ULN).
* History of hypersensitivity to study intervention or any excipients.
* History of any prior treatment with human growth hormone or related products (including insulin-like growth factor 1 [IGF-1]).
* History of receipt of any treatment that are known to potentially affect growth (including oral steroids >5 days in the last 6 months, high dose inhaled corticosteroids (>800 mcg/day beclametasone equivalent) and medication for attention deficit hyperactivity disorder).
* History of limb lengthening surgery (defined as distraction osteogenesis/Ilizarov/callostasis technique following submetaphyseal osteotomy to extend bone length).
* Any limb lengthening/corrective orthopaedic surgery planned at any point during the trial period.
* Less than 6 months since fracture or surgical procedure of any bone determined from the screening visit date.
* Presence of any internal guided growth plates/devices.
* History of removal of internal guided growth plates/devices within less than 6 months.
* History of receipt of any investigational product for achondroplasia or that may affect growth/interpretation of growth parameters.
* History of receipt of an investigational product (not for achondroplasia/growth affecting) within the last 30 days or 5 half-lives (whichever is longer).

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (6):
  - Ocean Sleep Medicine, Aliso Viejo, California
  - Ocean Sleep Medicine, Irvine, California
  - MemorialCare Sleep Disorders Center at Long Beach Memorial Medical Center, Long Beach, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Nemours Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Texas Children's Hospital, Houston, Texas
- Australia (2):
  - Murdoch Children's Research Institute, Melbourne, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitaire Ziekenhuizen Leuven (UZ Leuven), Leuven
- DanTrials ApS, Copenhagen NV, Denmark
- Fondazione Policlinico Universitario Agostino - Gemelli IRCCS, Roma, Italy
- Japan (2):
  - Osaka University Hospital, Suita, Osaka
  - Okayama University Hospital, Okayama
- Centro Hospitalar e Universitário de Coimbra - Hospital Pediátrico, Coimbra, Portugal
- Hospital Vithas San Jose, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4181005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 60 participants were enrolled, of which, 58 participants were assigned to treatment and 2 participants were not randomized, Out of 58 participants, 57 participants were treated. Note: The pharmacokinetics (PK) study cohort was not enrolled due to early study termination,
Groups:
- Recifercept 1 mg/kg QW: Children participants were enrolled and randomized to receive recifercept 1 mg/kg once weekly (QW) for 12 months.
- Recifercept 2 mg/kg BIW: Children participants were enrolled and randomized to receive recifercept 2 mg/kg twice weekly (BIW) for 12 months.
- Recifercept 1.5 mg/kg QD: Children participants were enrolled and randomized to receive recifercept 1.5 mg/kg once daily (QD) for 12 months.
Period: Overall Study
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Started (Assigned to treatment and treated) | 20 | 19 | 18
Completed | 16 | 17 | 3
Not Completed | 4 | 2 | 15
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1
Not completed — Study terminated by sponsor | 4 | 2 | 14

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least one dose of recifercept.
Groups:
- Total: Total of all reporting groups
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD | Total
Number analyzed (Participants) | 20 | 19 | 18 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.75 (2.84) | 5.16 (2.59) | 5.83 (2.31) | 5.58 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 6 | 24
  Male | 11 | 10 | 12 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 16 | 19 | 15 | 50
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 19 | 14 | 48
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study intervention in a participant who received study intervention. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. Relatedness to recifercept was assessed by the investigator (Yes/No).
Time Frame: The first dose up to 28 to 35 days after the last dose of study intervention (13 months)
Population: Analysis population included all participants who received at least 1 dose of recifercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Treatment-related AE | 7 | 15 | 14
  Treatment-related SAE | 0 | 0 | 0

2. Primary Outcome: Least Square Mean of Change From Baseline Height Growth at Month 3, Month 6, Month 9, and Month 12
Description: Height growth was defined as the ratio of observed change from baseline in standing height to the expected change from baseline in the reference population.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Ratio
  Month 3 | 1.1 [0.8 to 1.4] | 0.9 [0.6 to 1.2] | 0.6 [0.3 to 0.9]
  Month 6 | 0.9 [0.7 to 1.1] | 1.1 [0.9 to 1.3] | 1.0 [0.8 to 1.2]
  Month 9 | 1.0 [0.8 to 1.1] | 1.0 [0.8 to 1.1] | 1.0 [0.8 to 1.1]
  Month 12 | 1.0 [0.8 to 1.1] | 1.0 [0.9 to 1.1] | 0.9 [0.7 to 1.1]
Statistical Analysis 1: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; Results based on Mixed-Effect Repeated Measures (MMRM) analysis with gender as a covariate, participant (and/or time) as a random effect; treatment, visit, age and gender as fixed effects using an unstructured covariance matrix; Test type: Other; least square mean difference = 0.2, 95% CI 2-sided [-0.2 to 0.6] — Month 3
Statistical Analysis 2: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; Results based on MMRM analysis with gender as a covariate, participant (and/or time) as a random effect; treatment, visit, age and gender as fixed effects using an unstructured covariance matrix; Test type: Other; Least square mean difference = 0.5, 95% CI 2-sided [0.1 to 0.9] — Month 3
Statistical Analysis 3: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = -0.3, 95% CI 2-sided [-0.7 to 0.1] — Month 3
Statistical Analysis 4: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = -0.1, 95% CI 2-sided [-0.4 to 0.1] — Month 6
Statistical Analysis 5: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = -0.1, 95% CI 2-sided [-0.4 to 0.2] — Month 6
Statistical Analysis 6: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = -0.1, 95% CI 2-sided [-0.4 to 0.2] — Month 6
Statistical Analysis 7: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.2] — Month 9
Statistical Analysis 8: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.2] — Month 9
Statistical Analysis 9: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.2] — Month 9
Statistical Analysis 10: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = -0.0, 95% CI 2-sided [-0.2 to 0.2] — Month 12
Statistical Analysis 11: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-0.2 to 0.3] — Month 12
Statistical Analysis 12: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 2, analysis 2]; Test type: Other; Least square mean difference = -0.1, 95% CI 2-sided [-0.4 to 0.1] — Month 12

3. Secondary Outcome: Change From Baseline in Pulse Rate at Month 3, Month 6, Month 9, and Month 12
Description: Pulse rate measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (eg, television, cell phones) where possible (with consideration of the age of the child). Pulse rate was summarized by treatment in accordance with the sponsor reporting standards.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept. The "Number Analyzed" in a row was based on actual analyzed participants at each visit.
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
beats per minute (BPM)
  Baseline | 96.40 (16.583) | 97.58 (21.823) | 94.50 (15.497)
  Change at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Change at Month 3 | -1.47 (13.639) | -6.05 (20.871) | -2.94 (16.913)
  Change at Month 6: number analyzed (Participants) | 17 | 18 | 15
  Change at Month 6 | -2.65 (8.760) | -1.44 (15.659) | -2.20 (15.880)
  Change at Month 9: number analyzed (Participants) | 17 | 17 | 10
  Change at Month 9 | -4.35 (16.035) | -2.18 (17.746) | -15.20 (14.853)
  Change at Month 12: number analyzed (Participants) | 6 | 8 | 2
  Change at Month 12 | 1.17 (15.484) | -0.75 (34.012) | -11.50 (37.477)

4. Secondary Outcome: Change From Baseline in Respiratory Rate at Month 3, Month 6, Month 9, and Month 12
Description: Respiratory rate was obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Respiratory rate was summarized by treatment in accordance with the sponsor reporting standards.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
breaths/min
  Baseline | 23.15 (4.603) | 24.37 (3.905) | 23.39 (5.863)
  Change at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Change at Month 3 | 0.47 (5.691) | -1.00 (2.809) | -1.53 (4.939)
  Change at Month 6: number analyzed (Participants) | 17 | 18 | 15
  Change at Month 6 | -1.12 (3.516) | -0.94 (4.221) | 0.53 (4.502)
  Change at Month 9: number analyzed (Participants) | 17 | 17 | 10
  Change at Month 9 | -1.06 (3.473) | -0.94 (4.507) | -1.30 (6.945)
  Change at Month 12: number analyzed (Participants) | 7 | 8 | 2
  Change at Month 12 | 2.00 (5.132) | -3.75 (4.979) | 2.00 (15.556)

5. Secondary Outcome: Change From Baseline in Blood Pressure at Month 3, Month 6, Month 9, and Month 12
Description: Blood pressure measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (eg, television, cell phones) where possible (with consideration of the age of the child). Supine systolic blood pressure (SBP) and diastolic blood pressure (DBP) were summarized by treatment in accordance with the sponsor reporting standards.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
millimeters of mercury (mm Hg)
  Baseline (Supine DBP) | 66.55 (9.870) | 67.05 (9.897) | 62.11 (13.244)
  Change at Month 3 (Supine DBP): number analyzed (Participants) | 17 | 19 | 17
  Change at Month 3 (Supine DBP) | -0.76 (12.179) | -4.47 (8.618) | -0.29 (12.849)
  Change at Month 6 (Supine DBP): number analyzed (Participants) | 17 | 18 | 15
  Change at Month 6 (Supine DBP) | -3.65 (14.845) | -0.83 (10.837) | 5.27 (12.920)
  Change at Month 9 (Supine DBP): number analyzed (Participants) | 17 | 16 | 9
  Change at Month 9 (Supine DBP) | -3.41 (12.846) | -2.50 (11.408) | -2.44 (13.492)
  Change at Month 12 (Supine DBP): number analyzed (Participants) | 7 | 8 | 2
  Change at Month 12 (Supine DBP) | -3.14 (16.385) | -1.13 (13.953) | -4.50 (21.920)
  Baseline (Supine SBP) | 105.70 (10.732) | 118.37 (22.056) | 106.28 (14.199)
  Change at Month 3 (Supine SBP): number analyzed (Participants) | 17 | 19 | 17
  Change at Month 3 (Supine SBP) | 10.47 (14.261) | -5.68 (21.445) | 4.82 (15.134)
  Change at Month 6 (Supine SBP): number analyzed (Participants) | 17 | 18 | 15
  Change at Month 6 (Supine SBP) | 1.88 (21.863) | 3.94 (17.424) | 5.73 (14.587)
  Change at Month 9 (Supine SBP): number analyzed (Participants) | 17 | 16 | 9
  Change at Month 9 (Supine SBP) | 2.59 (15.732) | -2.94 (16.364) | 2.33 (19.371)
  Change at Month 12 (Supine SBP): number analyzed (Participants) | 7 | 8 | 2
  Change at Month 12 (Supine SBP) | 3.57 (27.700) | -11.75 (31.865) | -6.50 (4.950)

6. Secondary Outcome: Change From Baseline in Temperature at Month 3, Month 6, Month 9, and Month 12
Description: Temperature was obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Temperature measurements were summarized by treatment in accordance with the sponsor reporting standards.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degree Celsius (°C)
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Degree Celsius (°C)
  Baseline | 36.57 (0.441) | 36.43 (0.519) | 36.58 (0.466)
  Change at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Change at Month 3 | -0.06 (0.362) | -0.04 (0.297) | 0.11 (0.493)
  Change at Month 6: number analyzed (Participants) | 17 | 18 | 15
  Change at Month 6 | -0.08 (0.493) | -0.02 (0.298) | -0.03 (0.417)
  Change at Month 9: number analyzed (Participants) | 17 | 17 | 10
  Change at Month 9 | -0.16 (0.614) | -0.12 (0.437) | -0.20 (0.503)
  Change at Month 12: number analyzed (Participants) | 7 | 8 | 2
  Change at Month 12 | -0.21 (0.313) | -0.14 (0.316) | 0.30 (0.141)

7. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings at Month 3, Month 6, Month 9, and Month 12
Description: A physical examination included, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal systems and skin. Physical examination assessments were summarized by treatment in accordance with the sponsor reporting standards.
Time Frame: Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Abnormal Cardiovascular at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Abnormal Cardiovascular at Month 3 | 0 | 0 | 0
  Abnormal Cardiovascular at Month 6: number analyzed (Participants) | 17 | 19 | 15
  Abnormal Cardiovascular at Month 6 | 0 | 0 | 0
  Abnormal Cardiovascular at Month 9: number analyzed (Participants) | 16 | 17 | 9
  Abnormal Cardiovascular at Month 9 | 0 | 0 | 0
  Abnormal Cardiovascular at Month 12: number analyzed (Participants) | 16 | 16 | 3
  Abnormal Cardiovascular at Month 12 | 0 | 0 | 0
  Abnormal Gastrointestinal at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Abnormal Gastrointestinal at Month 3 | 0 | 0 | 0
  Abnormal Gastrointestinal at Month 6: number analyzed (Participants) | 17 | 19 | 15
  Abnormal Gastrointestinal at Month 6 | 0 | 1 | 0
  Abnormal Gastrointestinal at Month 9: number analyzed (Participants) | 16 | 17 | 9
  Abnormal Gastrointestinal at Month 9 | 0 | 2 | 0
  Abnormal Gastrointestinal at Month 12: number analyzed (Participants) | 16 | 16 | 3
  Abnormal Gastrointestinal at Month 12 | 0 | 0 | 0
  Abnormal Lungs at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Abnormal Lungs at Month 3 | 0 | 0 | 0
  Abnormal Lungs at Month 6: number analyzed (Participants) | 17 | 19 | 15
  Abnormal Lungs at Month 6 | 0 | 2 | 0
  Abnormal Lungs at Month 9: number analyzed (Participants) | 16 | 17 | 9
  Abnormal Lungs at Month 9 | 0 | 0 | 0
  Abnormal Lungs at Month 12: number analyzed (Participants) | 16 | 16 | 3
  Abnormal Lungs at Month 12 | 1 | 0 | 0
  Abnormal Skin at Month 3: number analyzed (Participants) | 17 | 19 | 17
  Abnormal Skin at Month 3 | 2 | 3 | 1
  Abnormal Skin at Month 6: number analyzed (Participants) | 17 | 19 | 15
  Abnormal Skin at Month 6 | 1 | 4 | 2
  Abnormal Skin at Month 9: number analyzed (Participants) | 16 | 17 | 9
  Abnormal Skin at Month 9 | 3 | 3 | 2
  Abnormal Skin at Month 12: number analyzed (Participants) | 16 | 16 | 3
  Abnormal Skin at Month 12 | 2 | 3 | 1

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Participants with laboratory abnormalities that met pre-specified criteria included following parameters: hematology (corpuscular volume, corpuscular hemoglobin, corpuscular hemoglobin concentration, platelet, leukocytes, lymphocytes, neutrophils, eosinophils, and monocytes), and chemistry (bilirubin, alkaline phosphatase, albumin, urea nitrogen, urate, potassium, phosphate, bicarbonate).
Time Frame: Baseline to Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Ery. Mean Corpuscular Volume (fL) < 0.9 x lower limit of normal (LLN) | 0 | 1 | 2
  Ery. Mean Corpuscular Volume (fL) > 1.1 x upper limit of normal (ULN) | 1 | 0 | 0
  Ery. Mean Corpuscular Hemoglobin (pg/cell) < 0.9 x LLN | 0 | 1 | 2
  Ery. Mean Corpuscular Hemoglobin Concentration (g/dL) < 0.9x LLN | 0 | 1 | 1
  Platelets (10^9/L) > 1.75 x ULN | 0 | 0 | 1
  Leukocytes (10^9/L) < 0.6 x LLN | 1 | 0 | 0
  Lymphocytes (10^9/L) < 0.8 x LLN | 5 | 9 | 4
  Neutrophils (10^9/L) < 0.8x LLN | 1 | 0 | 0
  Neutrophils (10^9/L) > 1.2 x ULN | 1 | 0 | 1
  Eosinophils (10^9/L) > 1.2 x ULN | 1 | 4 | 3
  Monocytes (10^9/L) > 1.2 x ULN | 4 | 1 | 1
  Bilirubin (mg/dL) > 1.5 x ULN | 0 | 1 | 0
  Alkaline Phosphatase (U/L) > 3.0 x ULN | 1 | 0 | 0
  Albumin (g/dL) > 1.2 x ULN | 2 | 3 | 1
  Urea Nitrogen (mg/dL) > 1.3 x ULN | 2 | 5 | 0
  Urate (mg/dL) > 1.2 x ULN | 2 | 1 | 0
  Potassium (mEq/L) > 1.1 x ULN | 2 | 4 | 4
  Phosphate (mg/dL) < 0.8 x LLN | 0 | 0 | 1
  Bicarbonate (mEq/L) < 0.9 x LLN | 2 | 2 | 4

9. Secondary Outcome: Pre-Dose Serum Concentration (Ctrough) of Recifercept
Description: Ctrough was defined as pre-dose serum concentration during dosing and observed directly from data.
Time Frame: Pre-dose on Day(s) 4, 8, 15, 29, 61, 91, 183, 273, 365
Population: Analysis population included all participants who received at least 1 dose of recifercept and had at least one evaluable concentration. The "Number Analyzed" in a row was based on actual analyzed participants at each visit.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
nanograms per millilitre (ng/mL)
  Day 4: number analyzed (Participants) | 18 | 19 | 16
  Day 4 | 215.8 (63.28) | 517.3 (174.18) | 1785.2 (651.92)
  Day 8: number analyzed (Participants) | 19 | 19 | 18
  Day 8 | 95.3 (23.35) | 614.6 (228.35) | 2682.6 (912.79)
  Day 15: number analyzed (Participants) | 18 | 19 | 17
  Day 15 | 137.1 (39.26) | 868.1 (341.98) | 3199.4 (1311.65)
  Day 29: number analyzed (Participants) | 17 | 19 | 16
  Day 29 | 154.3 (46.91) | 940.8 (415.45) | 3804.4 (1573.91)
  Day 61: number analyzed (Participants) | 17 | 19 | 17
  Day 61 | 183.8 (75.76) | 974.8 (604.47) | 3431.4 (1477.48)
  Day 91: number analyzed (Participants) | 17 | 19 | 15
  Day 91 | 225.5 (90.91) | 944.8 (466.38) | 3702.3 (2074.64)
  Day 183: number analyzed (Participants) | 17 | 19 | 15
  Day 183 | 370.9 (424.80) | 1078.9 (563.83) | 5185.5 (3190.30)
  Day 273: number analyzed (Participants) | 15 | 16 | 9
  Day 273 | 278.2 (140.41) | 1340.8 (695.10) | 3879.6 (3027.59)
  Day 365: number analyzed (Participants) | 15 | 16 | 3
  Day 365 | 249.5 (174.54) | 1320.4 (662.18) | 6766.7 (3145.18)

10. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) and Neutralizing Antibody (NAb) of Recifercept
Description: The immunogenicity was measured by presence of ADA and NAb in participants treated with recifercept and summarized by dose regimen.
Time Frame: The first dose up to 28 to 35 days after the last dose of study intervention (13 months)
Population: Analysis population included all participants who received at least 1 dose of recifercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Participants
  Overall incidence of positive ADA | 16 | 18 | 17
  Overall incidence of positive NAb | 13 | 16 | 16

11. Secondary Outcome: Change From Baseline in Sitting/Standing Height Ratio at Month 3, Month 6, Month 9, and Month 12
Description: Sitting/standing height ratio was the ratio of sitting height to standing height.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept. The "Overall Number of Participants Analyzed" was based on age 2-10 years at baseline. The "Number Analyzed" in a row was based on actual analyzed participants at each visit.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 18 | 18 | 18
Ratio
  Baseline: number analyzed (Participants) | 18 | 17 | 18
  Baseline | 0.7 (0.02) | 0.7 (0.02) | 0.7 (0.02)
  Change at Month 3: number analyzed (Participants) | 15 | 17 | 17
  Change at Month 3 | 0.0 (0.01) | -0.0 (0.01) | 0.0 (0.01)
  Change at Month 6: number analyzed (Participants) | 16 | 16 | 15
  Change at Month 6 | 0.0 (0.01) | -0.0 (0.01) | -0.0 (0.01)
  Change at Month 9: number analyzed (Participants) | 16 | 15 | 11
  Change at Month 9 | -0.0 (0.01) | -0.0 (0.01) | -0.0 (0.01)
  Change at Month 12: number analyzed (Participants) | 7 | 9 | 2
  Change at Month 12 | -0.0 (0.01) | -0.0 (0.01) | 0.0 (0.00)

12. Secondary Outcome: Least Square Mean of Change From Baseline Arm Span to Standing Height/Length Difference at Month 3, Month 6, Month 9, and Month 12
Description: Arm span to standing height/length difference was the difference between arm span and standing height.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept.
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeter (cm)
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
centimeter (cm)
  Month 3 | 0.4 [-0.2 to 1.0] | 0.0 [-0.5 to 0.6] | -0.6 [-1.2 to -0.0]
  Month 6 | 0.2 [-0.6 to 1.0] | 0.7 [-0.1 to 1.5] | -0.5 [-1.3 to 0.3]
  Month 9 | 0.7 [0.1 to 1.2] | 0.7 [0.2 to 1.2] | 0.0 [-0.6 to 0.6]
  Month 12 | 1.0 [-0.0 to 2.1] | 0.9 [-0.0 to 1.9] | 0.3 [-1.4 to 2.1]
Statistical Analysis 1: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; Results based on MMRM analysis with gender as a covariate, participant (and/or time) as a random effect; treatment, visit, treatment-by-visit interaction, age and gender as fixed effects using an unstructured covariance matrix; Test type: Other; Least square mean difference = 0.3, 95% CI 2-sided [-0.5 to 1.2] — Month 3
Statistical Analysis 2: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = 1.0, 95% CI 2-sided [0.2 to 1.8] — Month 3
Statistical Analysis 3: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = -0.7, 95% CI 2-sided [-1.5 to 0.1] — Month 3
Statistical Analysis 4: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = -0.5, 95% CI 2-sided [-1.6 to 0.6] — Month 6
Statistical Analysis 5: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = 0.7, 95% CI 2-sided [-0.4 to 1.9] — Month 6
Statistical Analysis 6: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = -1.2, 95% CI 2-sided [-2.3 to -0.1] — Month 6
Statistical Analysis 7: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = -0.0, 95% CI 2-sided [-0.8 to 0.7] — Month 9
Statistical Analysis 8: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = 0.6, 95% CI 2-sided [-0.2 to 1.5] — Month 9
Statistical Analysis 9: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = -0.7, 95% CI 2-sided [-1.5 to 0.2] — Month 9
Statistical Analysis 10: Comparison: Recifercept 1 mg/kg QW vs Recifercept 2 mg/kg BIW; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = 0.1, 95% CI 2-sided [-1.3 to 1.5] — Month 12
Statistical Analysis 11: Comparison: Recifercept 1 mg/kg QW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = 0.7, 95% CI 2-sided [-1.4 to 2.8] — Month 12
Statistical Analysis 12: Comparison: Recifercept 2 mg/kg BIW vs Recifercept 1.5 mg/kg QD; [analysis description as in outcome 12, analysis 1]; Test type: Other; Least square mean difference = -0.6, 95% CI 2-sided [-2.6 to 1.4] — Month 12

13. Secondary Outcome: Change From Baseline in Knee Height : Lower Segment Ratio at Month 3, Month 6, Month 9, and Month 12
Description: Knee height : lower segment ratio was the ratio of knee to heel length to the difference between standing height and sitting height.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Ratio
  Baseline: number analyzed (Participants) | 18 | 16 | 18
  Baseline | 0.81 (0.052) | 0.84 (0.058) | 0.80 (0.035)
  Change at Month 3: number analyzed (Participants) | 15 | 16 | 17
  Change at Month 3 | -0.00 (0.020) | -0.01 (0.052) | 0.02 (0.035)
  Change at Month 6: number analyzed (Participants) | 16 | 15 | 14
  Change at Month 6 | -0.00 (0.028) | -0.02 (0.062) | 0.00 (0.026)
  Change at Month 9: number analyzed (Participants) | 16 | 14 | 11
  Change at Month 9 | -0.00 (0.027) | -0.02 (0.065) | 0.01 (0.026)
  Change at Month 12: number analyzed (Participants) | 7 | 8 | 2
  Change at Month 12 | 0.00 (0.028) | -0.02 (0.081) | 0.02 (0.023)

14. Secondary Outcome: Change From Baseline in Occipito-Frontal Circumference at Month 3, Month 6, Month 9, and Month 12
Description: Head circumference or the occipito-frontal circumference is the greatest of the cranial dimensions which passes around the forehead anteriorly and the external occipital protruberance posteriorly. It is a routine part of the physical examination of a child and is of great importance in detecting abnormal patterns of cranial growth. Occipito-frontal circumference data were summarized for each treatment arm.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
cm
  Baseline: number analyzed (Participants) | 20 | 18 | 16
  Baseline | 54.56 (2.877) | 55.00 (2.179) | 56.13 (1.949)
  Change at Month 3: number analyzed (Participants) | 16 | 18 | 15
  Change at Month 3 | 0.19 (0.345) | 0.19 (0.382) | 0.30 (0.515)
  Change at Month 6: number analyzed (Participants) | 17 | 17 | 15
  Change at Month 6 | 0.33 (0.396) | 0.35 (0.506) | 0.30 (0.437)
  Change at Month 9: number analyzed (Participants) | 17 | 17 | 11
  Change at Month 9 | 0.46 (0.619) | 0.35 (0.597) | 0.54 (0.588)
  Change at Month 12: number analyzed (Participants) | 7 | 9 | 2
  Change at Month 12 | 0.87 (1.106) | 0.53 (0.557) | 0.00 (0.424)

15. Secondary Outcome: Change From Baseline in Occipito-Frontal to Occipito-Mid-Face Ratio at Month 3, Month 6, Month 9, and Month 12
Description: Ratio of occipito-frontal distance to occipito-mid-face measurements was summarized for each treatment arm.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Ratio
  Baseline: number analyzed (Participants) | 20 | 18 | 18
  Baseline | 1.00 (0.053) | 1.00 (0.055) | 1.00 (0.058)
  Change at Month 3: number analyzed (Participants) | 16 | 18 | 17
  Change at Month 3 | 0.01 (0.024) | 0.00 (0.039) | -0.01 (0.034)
  Change at Month 6: number analyzed (Participants) | 17 | 17 | 15
  Change at Month 6 | -0.01 (0.056) | 0.00 (0.027) | -0.02 (0.039)
  Change at Month 9: number analyzed (Participants) | 17 | 17 | 11
  Change at Month 9 | -0.01 (0.042) | -0.01 (0.034) | -0.02 (0.031)
  Change at Month 12: number analyzed (Participants) | 7 | 9 | 2
  Change at Month 12 | -0.04 (0.034) | -0.01 (0.028) | 0.00 (0.018)

16. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (Z-Score) at Month 3, Month 6, Month 9, and Month 12
Description: Height Standard Deviation Score (SDS) (z-score) was calculated as the difference between mean observed standing height at each visit and mean value of reference population divided by standard deviation of reference population. SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 18 | 18 | 18
SDS
  Baseline: number analyzed (Participants) | 18 | 17 | 18
  Baseline | -0.2 (0.91) | 0.1 (0.91) | 0.2 (1.26)
  Change at Month 3: number analyzed (Participants) | 15 | 17 | 17
  Change at Month 3 | 0.0 (0.13) | -0.0 (0.17) | 0.0 (0.26)
  Change at Month 6: number analyzed (Participants) | 16 | 16 | 15
  Change at Month 6 | 0.0 (0.21) | 0.0 (0.21) | 0.0 (0.24)
  Change at Month 9: number analyzed (Participants) | 16 | 16 | 11
  Change at Month 9 | 0.0 (0.26) | 0.0 (0.21) | 0.0 (0.20)
  Change at Month 12: number analyzed (Participants) | 7 | 9 | 2
  Change at Month 12 | 0.0 (0.33) | 0.1 (0.26) | -0.2 (0.17)

17. Secondary Outcome: Change From Baseline in Fixed Flexion Angles at Elbow at Month 3, Month 6, Month 9, and Month 12
Description: Fixed flexion angles at elbow data were presented for each treatment arm. An average of a participant's elbow extension measurements over a visit was computed.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees (°)
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
degrees (°)
  Baseline: number analyzed (Participants) | 20 | 18 | 16
  Baseline | -11.33 (20.002) | -18.31 (12.707) | -6.45 (17.628)
  Change at Month 3: number analyzed (Participants) | 16 | 18 | 14
  Change at Month 3 | 2.23 (8.976) | 4.29 (10.519) | 1.09 (5.285)
  Change at Month 6: number analyzed (Participants) | 16 | 17 | 14
  Change at Month 6 | -0.02 (16.407) | 2.80 (6.842) | 0.83 (5.742)
  Change at Month 9: number analyzed (Participants) | 17 | 17 | 11
  Change at Month 9 | -0.03 (16.659) | 4.83 (7.658) | 0.77 (10.621)
  Change at Month 12: number analyzed (Participants) | 7 | 9 | 2
  Change at Month 12 | 2.78 (34.075) | 1.00 (7.016) | -0.08 (0.825)

18. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 3, Month 6, Month 9, and Month 12
Description: Body Mass Index (BMI) = Weight (kg)/[(Standing Height (m))^2]. Standing height and weight were averaged over a visit before BMI was computed.
Time Frame: Baseline, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
kg/m^2
  Baseline: number analyzed (Participants) | 17 | 17 | 18
  Baseline | 19.83 (1.022) | 20.18 (1.318) | 21.57 (2.566)
  Change at Month 3: number analyzed (Participants) | 15 | 17 | 17
  Change at Month 3 | 0.10 (0.376) | -0.13 (0.400) | -0.01 (0.635)
  Change at Month 6: number analyzed (Participants) | 15 | 16 | 14
  Change at Month 6 | 0.25 (0.547) | 0.04 (0.500) | -0.21 (0.843)
  Change at Month 9: number analyzed (Participants) | 15 | 15 | 11
  Change at Month 9 | 0.36 (0.565) | 0.06 (0.593) | 0.02 (0.996)
  Change at Month 12: number analyzed (Participants) | 6 | 9 | 2
  Change at Month 12 | 0.12 (0.671) | -0.28 (0.569) | -0.50 (0.735)

19. Secondary Outcome: Change From Baseline in Waist : Chest Circumference Ratio at Month 9 and Month 12
Description: Waist : Chest Ratio = Waist Circumference / Chest Circumference. Waist and chest circumference were averaged over a visit before waist : chest circumference ratio was computed.
Time Frame: Baseline, Month 9, and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 20 | 19 | 18
Ratio
  Baseline: number analyzed (Participants) | 19 | 17 | 16
  Baseline | 0.93 (0.048) | 0.94 (0.051) | 0.97 (0.052)
  Change at Month 9: number analyzed (Participants) | 1 | 1 | 1
  Change at Month 9 | 0.07 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). | 0.00 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). | -0.01 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed).
  Change at Month 12: number analyzed (Participants) | 6 | 9 | 2
  Change at Month 12 | 0.05 (0.074) | 0.00 (0.063) | -0.01 (0.007)

20. Secondary Outcome: Change From Baseline in Apnea-Hypopnea Index (AHI) at Month 12
Description: The apnea-hypopnea index (AHI) is the average of the apneic and hypopneic episodes per hour of sleep, which is measured to assess obstructive sleep apnea (OSA). An AHI score of 1 to 4.9 events/hour is mild OSA, 5 to 9.9 events/hour is moderate, and more than 9 events/hour is severe in pediatric population.
Time Frame: Baseline and Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept and with a documented current diagnosis of sleep disordered breathing at enrollment. The "Number Analyzed" in a row was based on actual analyzed participants at each visit.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 7 | 4 | 8
events per hour
  Baseline (obstructive AHI) | 3.79 (4.720) | 1.20 (1.080) | 6.23 (6.881)
  Baseline (total AHI) | 6.34 (5.837) | 2.25 (2.872) | 16.07 (26.299)
  Change at Month 12 (obstructive AHI): number analyzed (Participants) | 3 | 1 | 0
  Change at Month 12 (obstructive AHI) | 0.31 (9.902) | -1.90 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). |
  Change at Month 12 (total AHI): number analyzed (Participants) | 3 | 1 | 0
  Change at Month 12 (total AHI) | -1.03 (8.671) | -2.90 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). |

21. Secondary Outcome: Change From Baseline in Desaturation Index at Month 12
Description: Desaturation index is one of the polysomnography parameters to assess obstructive sleep apnea. It refers to the average number of desaturation episodes occurring per hour, where desaturation episodes are defined as a decrease in the mean oxygen saturation of ≥3% (over the last 120 seconds) that lasts for at least 10 seconds.
Time Frame: Baseline and Month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: desaturations per hour
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 7 | 4 | 8
desaturations per hour
  Baseline | 4.90 (8.601) | 2.18 (2.502) | 13.53 (21.364)
  Change at Month 12: number analyzed (Participants) | 3 | 1 | 0
  Change at Month 12 | -4.61 (14.598) | 0.20 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). |

22. Secondary Outcome: Change From Baseline in Polysomnography Other Parameters at Month 12
Description: Polysomnography refers to a systematic process used to collect physiologic parameters during sleep. Polysomnography other parameters included total sleep time spent with oxygen saturation (SaO2) < 90% (T90), total sleep time spent with end-tidal carbon dioxide (EtCO2) >50 mm Hg.
Time Frame: Baseline and Month 12
Population: Analysis population included all participants who received at least 1 dose of recifercept and with a documented diagnosis of sleep-disordered breathing at enrollment. The "Number Analyzed" in a row was based on actual analyzed participants at each visit.
Measure: Mean (Standard Deviation); unit: percentage (%) of total sleep time
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 7 | 4 | 8
percentage (%) of total sleep time
  Baseline (T90): number analyzed (Participants) | 6 | 4 | 8
  Baseline (T90) | 16.43 (40.155) | 24.79 (49.472) | 0.72 (0.758)
  Change at Month 12 (T90): number analyzed (Participants) | 2 | 1 | 0
  Change at Month 12 (T90) | -48.95 (69.933) | -99.00 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). |
  Baseline (EtCO2): number analyzed (Participants) | 4 | 4 | 8
  Baseline (EtCO2) | 7.02 (14.030) | 9.50 (19.000) | 7.37 (17.355)
  Change at Month 12 (EtCO2): number analyzed (Participants) | 2 | 1 | 0
  Change at Month 12 (EtCO2) | -14.03 (19.841) | -38.00 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). |

23. Secondary Outcome: Change From Baseline in SaO2 Nadir at Month 12
Description: SaO2 measures the percentage of oxyhemoglobin (oxygen-bound hemoglobin) in the blood. SaO2 nadir refers to lowest SaO2.
Time Frame: Baseline and Month 12
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percentage (%) of oxyhemoglobin
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
Number analyzed (Participants) | 7 | 4 | 8
percentage (%) of oxyhemoglobin
  Baseline | 92.29 (3.147) | 94.25 (6.397) | 91.06 (5.882)
  Change at Month 12: number analyzed (Participants) | 3 | 1 | 0
  Change at Month 12 | -2.67 (7.095) | 1.00 (NA) — No summary statistics were provided for N <3 considering the insufficient number of participants (only 1 participant analyzed). |

ADVERSE EVENTS:
Time Frame: The first dose up to 28 to 35 days after the last dose of study intervention (13 months).
Arm/Group | Recifercept 1 mg/kg QW | Recifercept 2 mg/kg BIW | Recifercept 1.5 mg/kg QD
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 16/20 | 19/19 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recifercept 1 mg/kg QW (N=20) | Recifercept 2 mg/kg BIW (N=19) | Recifercept 1.5 mg/kg QD (N=18)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recifercept 1 mg/kg QW (N=20) | Recifercept 2 mg/kg BIW (N=19) | Recifercept 1.5 mg/kg QD (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 2 (2) | 3 (3)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 1 (5) | 0 (0) | 2 (3)
Injection site erythema (General disorders) | 4 (30) | 5 (17) | 4 (11)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (4) | 2 (2)
Injection site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (5) | 1 (2)
Injection site mass (General disorders) | 0 (0) | 1 (3) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 3 (3) | 3 (8) | 2 (9)
Injection site rash (General disorders) | 4 (7) | 4 (12) | 2 (5)
Injection site reaction (General disorders) | 0 (0) | 3 (5) | 1 (3)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 2 (4)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (3)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (4) | 3 (5) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 3 (4) | 2 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Impetigo (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (6) | 5 (7) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Otitis media (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Otitis media bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (5) | 1 (2)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood albumin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 3 (3) | 7 (7) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (5) | 1 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 2 (3) | 2 (8)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Antisocial behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (5)

LIMITATIONS AND CAVEATS:
The PK study cohort was not enrolled due to early study termination, therefore, the data of the PK cohort were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT04638153/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04638153/SAP_001.pdf